CLINICAL TRIAL: NCT00827645
Title: Effect of Uterine Artery Embolization on Symptoms of Pelvic Floor Dysfunction
Brief Title: Uterine Artery Embolization and Pelvic Floor Symptoms
Status: Withdrawn | Type: Observational
Why Stopped: never funded and never started
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 112008-033
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Leiomyoma; Incontinence; Prolapse
MeSH Terms: conditions — Leiomyoma; Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uterine artery embolization: Women with symptomatic uterine fibroids scheduled for uterine artery embolization

SUMMARY:
The objective of this study is to determine whether women who are already receiving treatment for their fibroids (ie. UAE) demonstrate improvement in urinary symptoms and sexual dysfunction as well.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 18-80 years
* symptomatic uterine fibroids
* scheduled for UAE
* Negative urine dipstick (negative result = trace or less for leukocytes & nitrites) or negative UA or negative culture (Urine dipstick is performed as standard of care)
* Available for 12-months of follow-up and able to complete study assessments, per clinician judgment
* Signed consent form

Exclusion Criteria:

* Age <18 or >80 years
* women who are unable to read and write English,
* pregnancy or planned pregnancy in the next 12 months
* < 6 months postpartum
* current use of anticholinergic medication, cholinergic agonists, tricyclic antidepressants, or duloxetine - must have been off such drugs for at least 4 weeks
* women with surgery for urinary incontinence or pelvic organ prolapse in the past 6 months
* history of bladder or pelvic cancer or pelvic radiation therapy
* prior augmentation cystoplasty
* urethral diverticulum, current or repaired.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with symptomatic uterine fibroids who are scheduled for uterine artery embolization
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Urinary symptoms as demonstrated by questionnaires | 1 year

SECONDARY OUTCOMES:
Sexual dysfunction as defined by questionnaires | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Y Wai, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States